CLINICAL TRIAL: NCT00807469
Title: Acute and Chronic Inflammatory Responses Induced by Smoking in Individuals Being Susceptible and Non-Susceptible for Development of COPD: From Specific Disease Phenotyping Towards Novel Made Therapy (Study 1)
Brief Title: Responses Induced by Smoking in Individuals Being Susceptible and Non-Susceptible for Development of COPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Top Institute Pharma (Other)
Collaborators: University Medical Center Groningen (Other); UMC Utrecht (Other); GlaxoSmithKline (Industry); Nycomed (Industry)
Responsible Party: Professor Dr DS Postma, Pulmonary Department UMCG Groningen, Postbus 9700 RB Groningen
Other Study IDs: 23440
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; smoking; susceptibility; inflammation; genetic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Disease Susceptibility; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be retained to investigate diffences in candidate genes (SNPs) for COPD between the 5 different groups.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- 1: 20 healthy individuals not susceptible for COPD (age 18-40 years, >0>10 packyears, FEV1/VC >70%, FEV1 >85% predicted)
- 2: 20 healthy individuals susceptible for COPD (age 18-40 years >20 packyears, FEV1/VC >70%, FEV1 >85% predicted) and high prevalence of COPD in smoking family members older than 45 years
- 3: 20 healthy individuals very susceptible for COPD (age 18-40 years, > 0 > 10 packyears, FEV1/VC >70%, FEV1 >85% predicted), and one of the smoking family members has severe early onset COPD or mild COPD with very low smoke exposure
- 4: 30 healthy individuals not susceptible for COPD (age 40-75 years, >20 packyears, FEV1/VC >70%, FEV1 >85% predicted)
- 5: 30 COPD patients with GOLD stage II (age 40-75 years, >10 packyears, FEV1/VC <_70%, FEV1 50-80% predicted)

SUMMARY:
COPD is ranked number 3 by the WHO list of important diseases worldwide and is the only disease with increasing mortality. The pathogenesis of cigarette smoke-induced COPD is obscure, therefore more insight is needed to design effective anti-inflammatory agents. We hypothesize that healthy individuals who are susceptible to smoking demonstrate a higher and aberrant inflammatory response to cigarette smoke. This susceptibility is caused by heterogeneous factors and is associated with various polymorphic genes that interact with each other and with the environment.

Objective:

* To define mediators involved in the early induction of COPD in susceptible smokers (and so to define new drug targets)
* To develop new biological and clinical markers for the early diagnosis and monitoring of COPD
* To compare between susceptible and non-susceptible individuals the corticosteroid responsiveness of bronchial epithelial cells in vitro, and to study the mechanisms of smoking-induced corticosteroid unresponsiveness.
* To study the role of candidate genes that may play a role in the development of fixed airway obstruction, and to identify clues for patient's responsiveness to specific drugs.

DETAILED DESCRIPTION:
Primary study parameters/outcome of the study:

* Local inflammation before and after cigarette smoking assessed by exhaled breath condensate, microprobe sampling and bronchial biopsies.
* Systemic inflammation before and after cigarette smoking assessed by the expression of established and newly developed markers on innate immune cells associated with pre-activation.
* Extensive clinical characterisation including life style factors, lung function, CT scanning of the lung.
* Corticosteroid responsiveness of epithelial cells in vitro.
* Distribution of candidate genes (SNPs) for COPD between the 5 different groups ( see description below) and associations with the inflammatory responses on acute smoking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Age, pack years, FEV1/FVC and FEV1% predicted must fit in one of the 5 groups described above.
* Able to stop smoking for 10 days and start smoking 3-4 cigarettes within 1 hour
* Physically and mentally able to undergo the total study protocol
* Written informed consent

Exclusion Criteria:

* Participation in another study
* Alpha-1-antitrypsin deficiency
* Selected grade 1-3 co-morbidity listed in the ACE-27
* Active pulmonary infection like tuberculosis, pneumonia, flue, tracheobronchitis
* Active extra-pulmonary infection like hepatitis A-C, cystitis, gastro-enteritis etc
* Pulmonary diseases like sarcoidosis, IPF, silicosis, hypersensitivity pneumonitis
* Life threatening diseases like carcinoma, AIDS (including HIV+), acute leukaemia etc
* Medication that may affect the results of the study: NSAID's, immunosuppressive agents like prednisolon, metotrexate, azathioprine,Acenocoumarol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy individuals and COPD patients with GOLD stage II. For detailed describtion see studie cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Local inflammation before and after cigarette smoking assessed by exhaled breath condensate, microprobe sampling and bronchial biopsies.

SECONDARY OUTCOMES:
Systemic inflammation before and after cigarette smoking assessed by the expression of established and newly developed markers on innate immune cells associated with pre-activation.
Extensive clinical characterisation including life style factors, lung function, CT scanning of the lung.
Distribution of candidate genes (SNPs) for COPD within the study population and associations with the inflammatory responses on acute smoking

CONTACTS AND LOCATIONS:
Overall Officials: Dirkje Postma, Dr. Prof. MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- Universitair Medisch Centrum Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Boudewijn IM, Faiz A, Steiling K, van der Wiel E, Telenga ED, Hoonhorst SJM, Ten Hacken NHT, Brandsma CA, Kerstjens HAM, Timens W, Heijink IH, Jonker MR, de Bruin HG, Sebastiaan Vroegop J, Pasma HR, Boersma WG, Wielders P, van den Elshout F, Mansour K, Spira A, Lenburg ME, Guryev V, Postma DS, van den Berge M. Nasal gene expression differentiates COPD from controls and overlaps bronchial gene expression. Respir Res. 2017 Dec 21;18(1):213. doi: 10.1186/s12931-017-0696-5. PMID 29268739
- [Derived] Loi ALT, Hoonhorst S, van Aalst C, Langereis J, Kamp V, Sluis-Eising S, Ten Hacken N, Lammers JW, Koenderman L. Proteomic profiling of peripheral blood neutrophils identifies two inflammatory phenotypes in stable COPD patients. Respir Res. 2017 May 22;18(1):100. doi: 10.1186/s12931-017-0586-x. PMID 28532454
- [Derived] Hoonhorst SJ, Lo Tam Loi AT, Pouwels SD, Faiz A, Telenga ED, van den Berge M, Koenderman L, Lammers JW, Boezen HM, van Oosterhout AJ, Lodewijk ME, Timens W, Postma DS, Ten Hacken NH. Advanced glycation endproducts and their receptor in different body compartments in COPD. Respir Res. 2016 Apr 26;17:46. doi: 10.1186/s12931-016-0363-2. PMID 27117828
- [Derived] Hoonhorst SJ, Timens W, Koenderman L, Lo Tam Loi AT, Lammers JW, Boezen HM, van Oosterhout AJ, Postma DS, Ten Hacken NH. Increased activation of blood neutrophils after cigarette smoking in young individuals susceptible to COPD. Respir Res. 2014 Oct 10;15(1):121. doi: 10.1186/s12931-014-0121-2. PMID 25301367
- [Derived] Hoonhorst SJ, ten Hacken NH, Lo Tam Loi AT, Koenderman L, Lammers JW, Telenga ED, Boezen HM, van den Berge M, Postma DS. Lower corticosteroid skin blanching response is associated with severe COPD. PLoS One. 2014 Mar 12;9(3):e91788. doi: 10.1371/journal.pone.0091788. eCollection 2014. PMID 24622644
- [Derived] Lo Tam Loi AT, Hoonhorst SJ, Franciosi L, Bischoff R, Hoffmann RF, Heijink I, van Oosterhout AJ, Boezen HM, Timens W, Postma DS, Lammers JW, Koenderman L, Ten Hacken NH. Acute and chronic inflammatory responses induced by smoking in individuals susceptible and non-susceptible to development of COPD: from specific disease phenotyping towards novel therapy. Protocol of a cross-sectional study. BMJ Open. 2013 Feb 1;3(2):e002178. doi: 10.1136/bmjopen-2012-002178. Print 2013. PMID 23377993